CLINICAL TRIAL: NCT07346404
Title: Dynamic 82-Rb Positron Emission Tomography (PET) for the Grading of KIDney Carcinoma
Acronym: RUBIKID
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Naogen Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP231442; 2024-514085-39-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-19; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; Positron Emission Tomography; Rubidium-82; neovascularization
MeSH Terms: conditions — Carcinoma, Renal Cell; Neovascularization, Pathologic | interventions — Rubidium-82

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 82-Rubidium (Other): 82-Rb; 10 MBq/kg intravenous injection over 30-60 seconds using an automated injection; two injections (Minimal injected activity per injection: 740 MBq ; maximal injected activity per injection: 1480 MBq).
  Interventions: Drug: 82-Rb injection

INTERVENTIONS:
Drug: 82-Rb injection — Injection of 82-Rb for 82-Rb PET imaging

SUMMARY:
This is a pilot prospective longitudinal monocentric, non-comparative, nonrandomised, and non-controlled open study.

is to test whether the intensity of 82-Rb uptake on PET acquisitions is associated to the aggressiveness of RCC on histology (ISUP grades), i.e., to successfully identify high-grade (ISUP grades 3 and 4) vs. lowgrade (ISUP grades 1 and 2) RCC.

DETAILED DESCRIPTION:
Tumoral vascularization is an important prognostic marker in renal cell carcinomas (RCC). The evaluation of RCC is often complex before surgery as only a small peripheral segment of the tumor is obtained with biopsy and tend to underestimate the aggressiveness and grade of RCC. Accurate noninvasive evaluation of the aggressiveness of RCC could improve the characterization of tumors before surgery and help guide patient management. Radiolabeled water has demonstrated its interest for the quantification of the vascularization of renal tumors in Positron Emission Tomography (PET). The synthesis of radiolabeled water requires, however, an on-site cyclotron, which is available only in a limited number of hospitals. 82-Rb, a potassium analog and positron-emitting radiotracer, is taken up by myocardial and renal cells. 82-Rb has been used for more than 15 years in North America for the quantification of myocardial perfusion with PET. The solution of 82-Rb chloride is obtained from 82-Sr / 82-Rb radiopharmaceutical generators which have recently obtained a marketing authorization in Europe. These generators can be installed in nuclear medicine departments in hospitals. Myocardial perfusion flow can be precisely quantified by modelling tissue uptake of the tracer on dynamic acquisitions obtained during the intravenous administration of 82-Rb chloride. Our hypothesis is that 82-Rb uptake profile could help grade noninvasively the aggressiveness of renal tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Signed written informed consent
* French Social Security affiliation
* Patients with high suspicion of or confirmed RCC requiring surgical resection
* Kidney tumor diameter between 2 cm and 7 cm with clear cell imaging feature (hyper vascular lesion with contrast-enhancement similar to the renal cortex on CTA)
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patient under legal protection (guardianship)
* Contraindication to the PET-CT
* Contraindication to the injection of 82-Rb
* Participation in another interventional study involving human participants or being in the exclusion period at the end of a previous study involving human participants, if applicable
* Patient on SMA (state medical aid)
* Unilateral renal agenesis
* Multicystic renal dysplasia
* Hereditary forms of RCC as VHL, MET, FH and FLCN
* Bosniak 3 cysts
* Hypovascular lesions with enhancement inferior to the renal cortex in corticomedullary-phase images on CTA
* Exclusion of clear renal cell adenocarcinoma on biopsy
* Kidney tumors with high suspicion of extra-renal extension (cT3b, cT3c, cN+ or M+).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Classify the aggressiveness of RCC into low grade and high grade based on the 82-Rb uptake intensity in renal tumors on PET. | Up to three months after surgery
  Intensity of 82-Rb uptake in the tumor is calculated as the tumor to background ratio (ratio between SUV max in the tumor and the mean SUV in normal renal parenchyma).
  High grades are tumors classified as ISUP 3 and 4 on pathology and low grades tumors classified as ISUP 1 and 2 on pathology.

SECONDARY OUTCOMES:
Correlation between the renal perfusion flow and the degree of neoangiogenesis in the tumor. | Up to three months after surgery
  The renal perfusion flow is measured on 82-Rb-PET. It is the maximum tumor flux, measured in tumors and expressed as ml/mn/g.
  The degree of neoangiogenesis is the degree of tumor vascularization measured on immuno-histology (CD34 and VEGF immunostaining). This degree for CD34 is calculated as the maximum density among four regions for CD34. The same applies to VEGF.
Association between imaging biomarkers on 82-Rb-PET and the histological type of the tumor. | Up to three months after surgery
  The imaging biomarkers are: maximal tumoral 82-Rb uptake (K1), ratio between maximal tumoral and non-tumoral renal perfusion, ratio between maximal tumoral and non-tumoral Rubidium uptake, standard deviation of perfusion values in the tumor, Standard deviation of 82-Rb uptake in the tumor calculated from the 82-Rb-PET acquisitions.
Association between imaging biomarkers on 82-Rb-PET and tumor aggressiveness (ISUP grades) in patients with clear-cell renal adenocarcinomas. | Up to three months after surgery
  Imaging biomarkers are: maximal tumoral 82-Rb uptake (K1), ratio between maximal tumoral and non-tumoral renal perfusion, ratio between maximal tumoral and non-tumoral Rubidium uptake, standard deviation of perfusion values in the tumor, Standard deviation of 82-Rb uptake in the tumor calculated from the 82-Rb-PET acquisitions.
Correlation between 82-Rb uptake and the degree of neoangiogenesis in the tumor. | Up to three months after surgery
  Rubidium uptake measured on 82-Rb-PET and degree of tumor vascularization measured on immuno-histology (CD34 and VEGF immunostaining).
Correlation between the estimated residual renal function and the observed renal function change. | Up to three months after surgery
  Estimated residual renal function based on 82-Rb-PET before surgery and change of creatinine clearance between baseline (the day of the 82-Rb-PET imagine) and three months after surgery.
To compare the diagnostic performance of biopsy and 82-Rb-PET for the ISUP grading of clear cell renal adenocarcinomas against the final results of histology (gold standard) of the renal tumor. | Up to three months after surgery
  Percentage of patients reclassified according to the gold-standard (ISUP grade of clear-cell renal adenocarcinomas on pathology).
Safety and tolerance of 82-Rb | Up to 72 hours after the PET with injection of the radiopharmaceutical
  Serious adverse events related to 82-Rb.

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Olivier TIMSIT, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Fabrien HYAFIL, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP - hôpital européen Georges-Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. The founder could be involved in the decision. Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization. Processing of shared data must comply with European General Data Protection Regulation (GDPR).